CLINICAL TRIAL: NCT04200599
Title: Amniotomy and Early Oxytocin Infusion Versus Amniotomy and Delayed Oxytocin Infusion in Nulliparous Women: a Randomised Controlled Trial
Brief Title: Early Versus Delayed Oxytocin Infusion Following Amniotomy in Nulliparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Azrai Abu, Clinical Consultant, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPI/111/8/JEP-2015-022
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Delivery Delayed; Mode of Delivery; Post Partum Hemorrhage; Uterine Hyperstimulation
Keywords: primigravida; amniotomy,; immediate oxytocin; delayed oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early oxytocin Infusion (Experimental): labour augmentation with oxytocin was started early following amniotomy.
  Interventions: Other: duration of initiation of oxytocin
- Late oxytocin infusion (Active Comparator): oxytocin augmentation was delayed at two hours after amniotomny and this practice is currently being used as standard protocol in this hospital to manage women in labour.
  Interventions: Other: duration of initiation of oxytocin

INTERVENTIONS:
Other: duration of initiation of oxytocin — mode of delivery

SUMMARY:
In UKM Medical Centre (UKMMC), delayed oxytocin augmentation at two hours following amniotomy is the routine obstetric practice in spontaneous or induced labour with intact membranes. This practice may potentially cause prolonged labour, extended labour room occupancy and increased maternal exhaustion while no additional benefit can be gained. On the other hand, recommendation for early oxytocin augmentation poses a dilemma as the effectiveness and safety of this practice are still in doubt.

Given this background, the aim of this study was to compare the effect of early versus delay oxytocin infusion in achieving successful vaginal delivery among the low-risk nulliparous women in UKMMC. Besides, this study also compares the adverse maternal and neonatal outcomes between the two practices.

DETAILED DESCRIPTION:
This was a randomised controlled trial undertaken in the labour room of UKMMC for a period of eighteen months from August 2014 until February 2016. Eligible women who were admitted in spontaneous labour or for induction of labour were recruited. For women who underwent induction of labour, an interval of at least six hours following vaginal prostaglandin before recruitment was mandatory to avoid overlapping effect of prostaglandin and oxytocin. Upon enrolment, each patient was given a study explanation and written consent was obtained.

The randomisation sequence, either to the early oxytocin group or the delayed oxytocin group, was generated using the computer randomisation program in block of two. Allocation to either arm of treatment was determined by the sequential opening of sealed numbered envelopes.

In the first arm of early oxytocin group, labour augmentation with oxytocin was started early following artificial ruptured of membrane(ARM). In the second arm of delayed oxytocin group, oxytocin augmentation was delayed at two hours after ARM and this practice is currently being used as standard protocol in this hospital to manage women in labour. In both arms,the infusion rate was doubled every 30 minutes to a maximum of 48 mL/h or until four to five moderate contractions per 10 minutes were achieved at which point the infusion rate was maintained. Continuous fetal heart rate monitoring was maintained throughout the intrapartum period. Vaginal examination was performed at four hours after ARM as well as when clinically indicated ie. abnormal cardiotocography (CTG) and maternal desire to bear down. In the presence of abnormal CTG, either fetal blood sampling or expedited delivery was undertaken as per decided by the obstetrician in charge.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 36+0 to 41+6 weeks
* singleton pregnancies in cephalic presentation
* estimated fetal weight between 2.5 - 4.0 kg
* cervical dilatation of 4 cm with intact membranes
* normal fetal heart rate trace before artificial rupture of membranes

Exclusion Criteria:

* Women with significant medical (eg. heart disease, pre-eclampsia, diabetes with high dose insulin, retroviral disease)
* fetal abnormality (eg. fetal growth restriction or small for gestational age < 2.5 kg, suspected macrosomia > 4.0 kg, fetal anomaly)

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — all primigravida
Enrollment: 250 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Achieving vaginal delivery | through study completion, an average of 18 months
  number of normal vaginal delivery
Neonatal outcome | through study completion, an average of 18 months
  Apgar score

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad azrai abu, Principal Investigator — Department of Obstetrics and Gynecology, UKM Medical Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Betran AP, Merialdi M, Lauer JA, Bing-Shun W, Thomas J, Van Look P, Wagner M. Rates of caesarean section: analysis of global, regional and national estimates. Paediatr Perinat Epidemiol. 2007 Mar;21(2):98-113. doi: 10.1111/j.1365-3016.2007.00786.x. PMID 17302638
- [Result] Barber EL, Lundsberg LS, Belanger K, Pettker CM, Funai EF, Illuzzi JL. Indications contributing to the increasing cesarean delivery rate. Obstet Gynecol. 2011 Jul;118(1):29-38. doi: 10.1097/AOG.0b013e31821e5f65. PMID 21646928
- [Result] O'Driscoll K, Jackson RJ, Gallagher JT. Prevention of prolonged labour. Br Med J. 1969 May 24;2(5655):477-80. doi: 10.1136/bmj.2.5655.477. PMID 5771578
- [Result] Dencker A, Berg M, Bergqvist L, Ladfors L, Thorsen LS, Lilja H. Early versus delayed oxytocin augmentation in nulliparous women with prolonged labour--a randomised controlled trial. BJOG. 2009 Mar;116(4):530-6. doi: 10.1111/j.1471-0528.2008.01962.x. PMID 19250364
- [Result] Hinshaw K, Simpson S, Cummings S, Hildreth A, Thornton J. A randomised controlled trial of early versus delayed oxytocin augmentation to treat primary dysfunctional labour in nulliparous women. BJOG. 2008 Sep;115(10):1289-95; discussion 1295-6. doi: 10.1111/j.1471-0528.2008.01819.x. PMID 18715415
- [Result] Selo-Ojeme DO, Pisal P, Lawal O, Rogers C, Shah A, Sinha S. A randomised controlled trial of amniotomy and immediate oxytocin infusion versus amniotomy and delayed oxytocin infusion for induction of labour at term. Arch Gynecol Obstet. 2009 Jun;279(6):813-20. doi: 10.1007/s00404-008-0818-x. Epub 2008 Oct 29. PMID 18958483
- [Result] Wei SQ, Luo ZC, Xu H, Fraser WD. The effect of early oxytocin augmentation in labor: a meta-analysis. Obstet Gynecol. 2009 Sep;114(3):641-649. doi: 10.1097/AOG.0b013e3181b11cb8. PMID 19701046
- [Result] Bugg GJ, Siddiqui F, Thornton JG. Oxytocin versus no treatment or delayed treatment for slow progress in the first stage of spontaneous labour. Cochrane Database Syst Rev. 2013 Jun 23;2013(6):CD007123. doi: 10.1002/14651858.CD007123.pub3. PMID 23794255
- [Result] Tan PC, Soe MZ, Sulaiman S, Omar SZ. Immediate compared with delayed oxytocin after amniotomy labor induction in parous women: a randomized controlled trial. Obstet Gynecol. 2013 Feb;121(2 Pt 1):253-259. doi: 10.1097/AOG.0b013e31827e7fd9. PMID 23344273
- [Result] Delgado Nunes V, Gholitabar M, Sims JM, Bewley S; Guideline Development Group. Intrapartum care of healthy women and their babies: summary of updated NICE guidance. BMJ. 2014 Dec 3;349:g6886. doi: 10.1136/bmj.g6886. No abstract available. PMID 25472418
- [Result] Liston R, Sawchuck D, Young D. No. 197a-Fetal Health Surveillance: Antepartum Consensus Guideline. J Obstet Gynaecol Can. 2018 Apr;40(4):e251-e271. doi: 10.1016/j.jogc.2018.02.007. PMID 29680082